CLINICAL TRIAL: NCT02593916
Title: Response to Medication Registry
Status: Completed | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 128024
Record Dates: First submitted 2015-10-29; First posted 2015-11-02 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Adverse Drug Events
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — * blood samples
  * buccal samples
Oversight: Data Monitoring Committee: No

SUMMARY:
To create a registry/database of patients who either have taken drugs that treat cardiovascular conditions or that have presented with cardiovascular symptoms that may be related to medication.

DETAILED DESCRIPTION:
To create a registry/database of patients who either have taken drugs that treat cardiovascular conditions or that have presented with cardiovascular symptoms that may be related to medication. Potential enrollees are those receiving (presently or in the past) the medicine(s) of interest. Subjects will be identified from computerized Intermountain Healthcare records. Patients receiving a drug of interest, both with and without an ADE will be enrolled in approximately equal numbers. Outpatients will be contacted by mail and invited to participate. Interested subjects will be instructed to return the enclosed response card with their intent indicated. The registry coordinator will contact interested subjects and the project will be explained. Willing participants will be enrolled either in person or via mail with the assistance of the project coordinator. Persons presenting in person for enrollment will be given the choice of venipuncture or buccal swab for sample collection for DNA extraction. In all cases informed consent will be obtained before collecting samples.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be > 18 years of age.
* The patient or legally authorized representative must sign a written informed consent, prior to sample collection, using a form that is approved by the local Institutional Review Board.
* The patient must have taken a medication of interest or have presented with a cardiovascular symptom possibly related to medication. The current medications of interest are as follows:

  * ACE inhibitors
  * ARBs
  * Aldosterone Antagonists
  * Alpha-Andrenergic Agonists
  * Anticoagulants
  * B-Type Natriuretic Peptides
  * Beta-blockers
  * Calcium Channel Blockers
  * Cardiac Glycosides
  * Antiarrhythmics
  * Combination Drugs
  * Diuretics
  * Electrolyte/Mineral Replacements
  * Lipid-lowering Medications
  * Positive Inotropes
  * Vasodilators/Nitrates
  * Statins
  * Antibiotics
  * Anthrocyclines

Exclusion Criteria:

* There are no exclusion criteria for this registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from existing Intermountain Healthcare databases and registries who either have taken drugs that treat cardiovascular conditions or that have presented with cardiovascular symptoms that may be related to medication.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2007-03; Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Genetic and biomarker correlates with clinical response(s) to medication | 5 years
  We will monitor clinical responses to medications for 5 years and look for genetic markers and biomarkers that correlate with these responses.

SECONDARY OUTCOMES:
Dosage adjustments | 5 years
  We will monitor medication dosage adjustments for 5 years and look for genetic markers and biomarkers that correlate with these adjustments.
Beneficial responses | 5 years
  We will monitor beneficial responses to medications for 5 years and look for genetic markers and biomarkers that correlate with these responses.
Adverse drug events | 5 years
  We will monitor adverse drug events for 5 years and look for genetic markers and biomarkers that correlate with these events.
Drug interactions | 5 years
  We will monitor drug interactions for 5 years and look for genetic markers and biomarkers that correlate with these interactions.

CONTACTS AND LOCATIONS:
Overall Officials: John F Carlquist, PhD, Principal Investigator — LDS Hospital
Locations (1):
- LDS Hospital, Salt Lake City, Utah, United States